CLINICAL TRIAL: NCT02135848
Title: A Multi-center, Placebo-controlled Study to Evaluate the Safety and Efficacy of GSK1278863 vs. Placebo in Subjects With Peripheral Artery Disease (PAD).
Brief Title: 3 Month PHI PAD PoM Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 114272
Record Dates: First submitted 2012-06-28; First posted 2014-05-12 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-08

CONDITIONS: Vascular Disease, Peripheral
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1278863 (Experimental): Study Drug
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863
  Arms: GSK1278863
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, blinded, placebo controlled study to evaluate the safety of GSK1278863 and its acute and short-term (e.g. 14d) effects on calf muscle endurance and walking ability in subjects with PAD and symptomatic claudication.

DETAILED DESCRIPTION:
This is a multi-center, randomized, blinded, placebo controlled study to evaluate the safety of GSK1278863 and its acute and short-term (e.g. 14d) effects on calf muscle endurance and walking ability in subjects with PAD and symptomatic claudication. Functional assessments will be performed following a single high dose (300mg), a single low dose (15mg), and following 14 days of low dose treatment (15mg q.d.). The objectives of this study are to: 1) Evaluate the safety and tolerability of GSK1278863 administered as a single dose and as sub-chronic low dosing (i.e. 14 days) in subjects with peripheral artery disease; 2) To demonstrate the potential pharmacodynamic effect of GSK1278863 on functional measures of calf muscle endurance and fatigability and timed walking distance following a single high or low dose and after 14 days of multiple low dose administration in subjects with claudication-limited peripheral artery disease. In this hypothesis-generating study, multiple assessments of ambulatory and skeletal muscle function will be made during standardized tests of claudication-limited exercise performance, and 3). Characterize the relationship, if any, between the doses and plasma concentrations of GSK1278863 and the pharmacodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 40 years of age.
* Male subjects must use one of the contraceptive methods listed in Section 8.1 for 90 days post-last dose.
* Females must be postmenopausal, surgically sterilized, or practicing a suitable method of birth control so that in the opinion of the investigator they will not become pregnant during the course of the study.

A female subject is eligible to participate if she is of child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 30 days post-last dose.

* Peripheral artery disease defined as an ankle-brachial index (ABI) at rest ≤ 0.90 in at least one leg in which the patient experiences claudication. For all subsequent evaluations, the Index Leg refers to the symptomatic leg with the lowest ABI.
* Claudication symptoms with stable severity for at least 3 months prior to screening.
* The patient is able to provide written informed consent to participate in this study.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin greater than or equal too 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Confirmed QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with bundle branch block.
* Subjects must be able to perform performance/exercise testing

Exclusion Criteria:

* Coronary artery bypass graft (CABG), open peripheral vascular procedures, or major surgical procedures within 6 months prior to screening or patients likely to require revascularization during the course of the trial. Endovascular procedures within 3 months prior to screening.
* Any unstable vascular syndromes (such as TIA, CVA, unstable angina or acute MI), including major changes to related medications, within 6 months prior to randomization.
* Critical leg ischemia classified as Fontaine Stage III-IV (rest pain, tissue necrosis or gangrene).
* Pregnant or nursing women (women capable of childbearing must have a negative pregnancy test).
* A hemoglobin value at screening is:

Male subjects or post-menopausal females: > 15.5 g/dL Female subjects: > 14.5 g/dL

* Active malignancy or diagnosis of malignancy within 5 years prior to screening (excluding successfully treated basal or squamous cell carcinoma).
* Other clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the Investigator or the Medical Monitor, not stabilized or may otherwise confound the results of the study.
* Patients with a baseline medical history of proliferative diabetic retinopathy, preproliferative diabetic retinopathy, or wet age-related macular degeneration (AMD)
* Previously enrolled in a gene therapy clinical study unless patient was randomized to placebo.
* Plans to initiate a formal exercise training program during the course of the study, or initiation of a formal exercise training program within 3 months prior to screening.
* Poorly controlled hypertension (defined as seated resting BP >160 mmHg systolic or > 95 mmHg diastolic, or both).
* Hypotension (defined as seated resting BP < 95 mmHg systolic or < 55 mmHg diastolic, or both, or symptomatic hypotension [seated, supine, or orthostatic]).
* Exercise tolerance, including bilateral heel raise and Six-Minute Walk Test performance, that is limited by co-morbid conditions or diseases other than claudication.
* Poorly controlled diabetes defined as Hemoglobin A1c (HbA1c) > 10%.
* Creatinine > 2.5 mg/dL or undergoing hemodialysis.
* Thrombocytopenia defined as platelet count < 100,000/mm3 at screening.
* Hematocrit ≤ 30% or ≥ 55%.
* International Normalized Ratio (INR) > 1.5.
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result if performed within 3 months of screening (testing not required at Screening).
* History of alcohol or drug abuse, or a significant medical or psychiatric disorder that may impair compliance with the requirements of the protocol.
* The patient has received an investigational drug within 30 days prior to this study.
* The patient is enrolled or plans to enroll in another clinical trial during this study
* History of venous thrombosis, defined as deep vein thrombosis, pulmonary embolism or other venous thrombotic condition, within 1 year prior to Screening.
* Acute peptic ulcer disease or history of chronic rectal bleeding.
* Patients with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue.
* Use of prescription drugs within 7 days prior to first dose of study drug (Day 1) until after completion of all study drug doses and Day 35 assessments:

which are known to be inhibitors of CYP 2C8 OR which are known to be both CYP 2C8 and OATP1B1 substrates OR which rely mainly on OATP1B1/1B3 for hepatic clearance as described in Section 9 of the protocol.

* Use of prescription drugs within 14 days prior to first dose of study drug (Day 1) until completion of all study drug doses and Day 35 assessments, which are known to be inducers of CYP 2C8, as described in Section 9 of the protocol.
* Use of non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug (Day 1) through the Follow-up Visit (Day 65), unless, in the opinion of the Investigator, medication will not interfere with the study procedures or compromise subject safety and GSK Medical Monitor concurs.
* History of sensitivity to any of the study drugs, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Patient is mentally or legally incapacitated.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10-15 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114272 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 centers in the United States from 15-October-2010 to 01-November-2011.
Groups:
- GSK1278863: Eligible participants received an initial single high dose of 300 milligram (mg) GSK1278863 tablets orally followed by a 14-day washout period. After completing the washout period, participants received repeated dose of 15 mg GSK1278863 tablets orally once daily for 14 days.
- Placebo: Eligible participants received single dose of placebo matched with 300 mg GSK1278863 tablets orally followed by a 14-day washout period. After completing the washout period, participants received placebo matched with 15 mg GSK1278863 tablets orally once daily for 14 days.
Period: Overall Study
Arm/Group | GSK1278863 | Placebo
Started | 26 | 20
Completed | 23 | 19
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1278863: Eligible participants received an initial single high dose of 300 mg GSK1278863 tablets orally followed by a 14-day washout period. After completing the washout period, participants received repeated dose of 15 mg GSK1278863 tablets orally once daily for 14 days.
- Total: Total of all reporting groups
Arm/Group | GSK1278863 | Placebo | Total
Number analyzed (Participants) | 26 | 20 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (9.50) | 69.4 (7.65) | 68.8 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 19 | 14 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 19 | 14 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 67 days
Population: Safety population which comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1278863 300 mg: Eligible participants received an initial single high dose of 300 mg GSK1278863 tablets orally.
- Placebo Matched With GSK1278863 300 mg: Eligible participants received single dose of placebo matched with 300 mg GSK1278863 tablets orally.
- GSK1278863 15 mg: Eligible participants received repeated dose of 15 mg GSK1278863 tablets orally once daily for 14 days.
- Placebo Matched With GSK1278863 15 mg: Eligible participants received placebo matched with 15 mg GSK1278863 tablets orally once daily for 14 days.
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
Number analyzed (Participants) | 26 | 20 | 23 | 19
Participants
  AE | 14 | 6 | 9 | 3
  SAE | 2 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were recorded with the participant lying supine, having rested in this position for at least 5 minutes before each recording. Full 12 lead ECGs were recorded using an ECG device that automatically calculated the heart rate and measured PR, QRS, RR, QT and QT, QT corrected by Bazett's formula (QTcB) and QT corrected by Fridericia's formula (QTcF) intervals. Number of participants with abnormal (not clinically significant [NCS] and clinically significant [CS]) ECG findings are presented.
Time Frame: Up to 39 days
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
Number analyzed (Participants) | 26 | 20 | 23 | 19
Participants
  Acute Day 1, Pre-dose; Abnormal NCS: number analyzed (Participants) | 26 | 20 | 0 | 0
  Acute Day 1, Pre-dose; Abnormal NCS | 14 | 16 |  |
  Acute Day 1, Pre-dose; Abnormal CS: number analyzed (Participants) | 26 | 20 | 0 | 0
  Acute Day 1, Pre-dose; Abnormal CS | 0 | 0 |  |
  Acute Day 1, 2.5 hour; Abnormal NCS: number analyzed (Participants) | 26 | 20 | 0 | 0
  Acute Day 1, 2.5 hour; Abnormal NCS | 15 | 14 |  |
  Acute Day 1, 2.5 hour; Abnormal CS: number analyzed (Participants) | 26 | 20 | 0 | 0
  Acute Day 1, 2.5 hour; Abnormal CS | 0 | 0 |  |
  Chronic Day 1, Pre-dose; Abnormal NCS: number analyzed (Participants) | 0 | 0 | 23 | 19
  Chronic Day 1, Pre-dose; Abnormal NCS |  |  | 12 | 14
  Chronic Day 1, Pre-dose; Abnormal CS: number analyzed (Participants) | 0 | 0 | 23 | 19
  Chronic Day 1, Pre-dose; Abnormal CS |  |  | 0 | 0
  Chronic Day 1, 2.5 hour; Abnormal NCS: number analyzed (Participants) | 0 | 0 | 23 | 19
  Chronic Day 1, 2.5 hour; Abnormal NCS |  |  | 8 | 14
  Chronic Day 1, 2.5 hour; Abnormal CS: number analyzed (Participants) | 0 | 0 | 23 | 19
  Chronic Day 1, 2.5 hour; Abnormal CS |  |  | 0 | 0
  End of treatment, Pre-dose; Abnormal NCS: number analyzed (Participants) | 0 | 0 | 23 | 19
  End of treatment, Pre-dose; Abnormal NCS |  |  | 15 | 14
  End of treatment, Pre-dose; Abnormal CS: number analyzed (Participants) | 0 | 0 | 23 | 19
  End of treatment, Pre-dose; Abnormal CS |  |  | 0 | 0
  Early termination, Pre-dose; Abnormal NCS: number analyzed (Participants) | 3 | 0 | 0 | 0
  Early termination, Pre-dose; Abnormal NCS | 2 |  |  |
  Early termination, Pre-dose; Abnormal CS: number analyzed (Participants) | 3 | 0 | 0 | 0
  Early termination, Pre-dose; Abnormal CS | 1 |  |  |

3. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital signs included heart rate, systolic and diastolic blood pressure and were performed with the participant in a supine position after the participant had rested for at least 5 minutes. Number of participants with vital signs of potential clinical importance are presented.
Time Frame: Up to 39 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
Number analyzed (Participants) | 26 | 20 | 23 | 19
Participants | 3 | 1 | 2 | 3

4. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: Clinical chemistry analyte of potential clinical concern included albumin, calcium, creatinine, glucose, magnesium, phosphorus, potassium, sodium and bicarbonate. Number of participants with clinical chemistry abnormalities of potential clinical importance are presented.
Time Frame: Up to 67 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
Number analyzed (Participants) | 26 | 20 | 23 | 19
Participants
  High Glucose | 5 | 2 | 5 | 3
  High Calcium | 0 | 0 | 1 | 0
  High Potassium | 1 | 1 | 2 | 1
  Low Carbon-dioxide content | 0 | 0 | 1 | 1
  High Creatinine | 1 | 0 | 1 | 0
  High Carbon-dioxide content | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Clinical Hematology Abnormalities of Potential Clinical Importance
Description: Hematology parameters included platelet count, red blood cell (RBC) count, white blood cell WBC count (absolute), hemoglobin, hematocrit, Mean corpuscular volume (MCV), Mean corpuscular hemoglobin (MCH), Mean corpuscular hemoglobin concentration (MCHC), neutrophils, lymphocytes, monocytes, eosinophils and basophils. Number of participants with clinical hematology abnormalities of potential clinical importance are presented.
Time Frame: Up to 67 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Eligible participants received placebo matched with 300 mg GSK1278863 tablets orally followed by a 14-day washout period. After completing the washout period, participants received placebo matched with 15 mg GSK1278863 tablets orally once daily for 14 days.
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Participants | 0 | 0

6. Secondary Outcome: Change From Baseline in Total Number of Contractions to Onset of Claudication
Description: At Visit 1 (-21 to -10 days), the participant was introduced to the bilateral heel raise test (BHRT). Test familiarization consisted of the participant performing heel raises to the onset of claudication. The BHRT was conducted with an electrogoniometer instrumented on the index leg. Successive heel raise repetitions were performed once every other second until the participant stopped due to intolerable claudication pain or fatigue, or other criteria for stopping the test were met. The index leg was defined as the leg that met the inclusion symptomatic and hemodynamic criteria (ankle brachial index [ABI] ≤ 0.90) with the lowest ABI considered if both legs were affected. Baseline was Day 1. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population comprised of all participants who provided pharmacodynamic data, i.e. bilateral heel-raise data or six-minute-walk-test data. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Contractions
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Contractions
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 2.52 (7.7) | -1.67 (6.5)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 22 | 18
  Acute Day 2, Pre-dose | 3.77 (8.6) | -0.94 (4.8)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 5.68 (10.0) | -1.56 (5.1)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 3.00 (9.4) | 0.83 (8.6)
  End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  End of treatment, Pre-dose | 2.90 (9.2) | -0.83 (6.4)

7. Secondary Outcome: Change From Baseline in Total Work Performed to Onset of Claudication
Description: BHRT is a method to assess muscle performance in participants with claudication. Participants with peripheral artery disease (PAD) and claudication experience reproducible symptoms of leg pain during walking exercise. The symptom of claudication is due to exercise-induced ischemia of muscles in legs, most commonly in calf muscles. At Visit 1 (-21 to -10 days), the participant was introduced to BHRT. Test familiarization consisted of the participant performing heel raises to onset of claudication. BHRT was conducted with an electrogoniometer instrumented on the index leg (leg that met the inclusion symptomatic and hemodynamic criteria [ABI ≤ 0.90] with the lowest ABI considered if both legs were affected). Successive heel raise repetitions were performed once every other second until participant stopped due to intolerable claudication pain/fatigue, or other criteria for stopping the test were met. Baseline was Day 1. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram-meters
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
kilogram-meters
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 14.66 (42.0) | -8.12 (52.5)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 22 | 18
  Acute Day 2, Pre-dose | 12.46 (42.5) | -14.61 (55.2)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 24.17 (38.7) | -15.69 (45.0)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 11.23 (40.6) | -3.03 (68.0)
  End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  End of treatment, Pre-dose | 8.13 (42.1) | -15.60 (59.1)

8. Secondary Outcome: Change From Baseline in Total Exercise Time to Onset of Claudication
Description: BHRT is a method to assess muscle performance in participants with claudication. Participants with PAD and claudication experience reproducible symptoms of leg pain during walking exercise. The symptom of claudication is due to exercise-induced ischemia of muscles in legs, most commonly in calf muscles. At Visit 1 (-21 to -10 days), the participant was introduced to the BHRT. Test familiarization consisted of the participant performing heel raises to the onset of claudication. The BHRT was conducted with an electrogoniometer instrumented on the index leg (the leg that met the inclusion symptomatic and hemodynamic criteria [ABI ≤ 0.90] with the lowest ABI considered if both legs were affected). Successive heel raise repetitions were performed once every other second until the participant stopped due to intolerable claudication pain or fatigue, or other criteria for stopping the test were met. Baseline was Day 1. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Seconds
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 4.39 (15.7) | -3.34 (13.4)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 22 | 18
  Acute Day 2, Pre-dose | 8.00 (17.2) | -3.96 (14.4)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 10.50 (19.9) | -3.71 (11.1)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 5.63 (18.5) | 1.25 (18.3)
  End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  End of treatment, Pre-dose | 5.03 (18.7) | -1.05 (11.8)

9. Secondary Outcome: Change From Baseline in Total Number of Contractions to Claudication-limited Maximal Muscle Performance
Description: as for outcome 8
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Contractions
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Contractions
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 1.00 (7.6) | -2.17 (6.4)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 23 | 18
  Acute Day 2, Pre-dose | 1.48 (10.1) | -0.94 (5.6)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 4.55 (8.3) | -1.83 (5.6)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 3.45 (10.0) | -0.67 (6.9)
  End of treatment, Pre-dose: number analyzed (Participants) | 22 | 18
  End of treatment, Pre-dose | 3.45 (10.1) | -1.11 (8.1)

10. Secondary Outcome: Change From Baseline in Total Work Performed to Claudication-limited Maximal Muscle Performance
Description: as for outcome 8
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram-meters
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
kilogram-meters
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 11.32 (46.1) | -6.20 (53.4)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 23 | 18
  Acute Day 2, Pre-dose | 5.11 (55.4) | -11.35 (62.2)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 22.20 (36.5) | -10.84 (62.3)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 14.40 (46.8) | -4.04 (68.9)
  End of treatment, Pre-dose: number analyzed (Participants) | 22 | 18
  End of treatment, Pre-dose | 6.75 (37.1) | -14.22 (75.6)

11. Secondary Outcome: Change From Baseline in Total Exercise Time to Claudication-limited Maximal Muscle Performance
Description: as for outcome 8
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
seconds
  Acute Day 1, 3 hour: number analyzed (Participants) | 25 | 18
  Acute Day 1, 3 hour | 0.15 (14.7) | -5.41 (13.3)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 23 | 18
  Acute Day 2, Pre-dose | 2.18 (21.1) | -5.06 (15.8)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 5.71 (15.7) | -4.91 (12.3)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 20 | 18
  Chronic Day 1, 3 hour | 4.89 (18.6) | -2.92 (15.2)
  End of treatment, Pre-dose: number analyzed (Participants) | 22 | 18
  End of treatment, Pre-dose | 4.59 (21.1) | -2.69 (15.7)

12. Secondary Outcome: Change From Baseline in the Maximal Distance Covered During a Six-Minute Walk Test
Description: The Six-Minute Walk Test was performed by the participant walking at a self-selected pace for 6 minutes through a pre-defined walking course. When the Six-Minute Walk Test and Bilateral Heel Raise Test were conducted at the same study visit, the participant was allowed to rest a minimum of one hour between these tests. Baseline was Day 1. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Feet
  Acute Day 1, 2 hour | -52.88 (140.3) | -11.60 (64.3)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 24 | 19
  Acute Day 2, Pre-dose | -42.25 (160.9) | -7.11 (116.2)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 23 | 19
  Chronic Day 1, Pre-dose | 8.43 (139.7) | -31.89 (138.6)
  Chronic Day 1, 2 hour: number analyzed (Participants) | 23 | 19
  Chronic Day 1, 2 hour | -6.43 (145.2) | -26.53 (166.6)
  End of treatment, Pre-dose: number analyzed (Participants) | 23 | 19
  End of treatment, Pre-dose | 14.57 (163.9) | -47.47 (192.8)

13. Secondary Outcome: Change From Baseline in Erythropoietin Concentration
Description: Blood samples for analysis of fasting levels of erythropoietin, was collected up to end of treatment or early termination. Baseline acute was Day 1 and Baseline chronic was Day 21. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Units per Liter
  Acute Day 1, 2.5 hour | 8.10 (14.119) | -2.54 (3.718)
  Acute Day 1, 3 hour | 53.98 (87.176) | -2.25 (4.416)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 18 | 19
  Acute Day 2, Pre-dose | 907.43 (561.105) | -0.79 (6.889)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 23 | 19
  Chronic Day 1, Pre-dose | -1.05 (8.228) | -2.39 (6.275)
  Chronic Day 1, 2.5 hour: number analyzed (Participants) | 23 | 18
  Chronic Day 1, 2.5 hour | -2.24 (7.349) | -5.18 (7.905)
  Chronic Day 1, 3 hour: number analyzed (Participants) | 23 | 18
  Chronic Day 1, 3 hour | 1.00 (8.435) | -4.81 (8.067)
  End of treatment, Pre-dose: number analyzed (Participants) | 23 | 19
  End of treatment, Pre-dose | 0.78 (11.360) | -1.60 (13.421)
  Early termination: number analyzed (Participants) | 2 | 0
  Early termination | -10.15 (7.283) |

14. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood samples for analysis of fasting levels of hemoglobin was collected up to end of treatment or early termination. Baseline acute was Day 1 and Baseline chronic was Day 21. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Grams per Liter
  Acute Day 2, Pre-dose: number analyzed (Participants) | 24 | 19
  Acute Day 2, Pre-dose | 1.29 (5.706) | -0.84 (5.776)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 20
  Chronic Day 1, Pre-dose | 0.91 (7.596) | -0.44 (5.973)
  End of treatment, Pre-dose: number analyzed (Participants) | 23 | 19
  End of treatment, Pre-dose | 9.13 (9.221) | -1.42 (5.470)
  Early termination: number analyzed (Participants) | 2 | 0
  Early termination | 2.50 (2.121) |
  Follow-up: number analyzed (Participants) | 25 | 18
  Follow-up | 6.36 (6.350) | -1.17 (7.786)

15. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples for analysis of fasting levels of hematocrit was collected up to end of treatment or early termination. Baseline acute was Day 1 and Baseline chronic was Day 21. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Fraction
  Acute Day 2, Pre-dose: number analyzed (Participants) | 24 | 19
  Acute Day 2, Pre-dose | 0.00 (0.017) | -0.00 (0.018)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 22 | 18
  Chronic Day 1, Pre-dose | 0.00 (0.021) | 0.00 (0.017)
  End of treatment, Pre-dose: number analyzed (Participants) | 23 | 19
  End of treatment, Pre-dose | 0.03 (0.029) | -0.00 (0.015)
  Early termination: number analyzed (Participants) | 2 | 0
  Early termination | 0.02 (0.002) |
  Follow-up: number analyzed (Participants) | 25 | 18
  Follow-up | 0.02 (0.023) | -0.00 (0.023)

16. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP)
Description: Blood samples for analysis of fasting levels of hsCRP, was collected up to end of treatment or early termination. Baseline acute was Day 1 and Baseline chronic was Day 21. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams/Liter (mg/L)
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Milligrams/Liter (mg/L)
  Acute Day 2, Pre-dose: number analyzed (Participants) | 23 | 16
  Acute Day 2, Pre-dose | 2.51 (1.905) | -0.08 (2.183)
  Chronic Day 1, Pre-dose: number analyzed (Participants) | 21 | 14
  Chronic Day 1, Pre-dose | 1.12 (2.909) | 0.21 (3.550)
  End of treatment, Pre-dose: number analyzed (Participants) | 21 | 15
  End of treatment, Pre-dose | 1.32 (3.467) | 0.72 (5.625)
  Early termination: number analyzed (Participants) | 2 | 0
  Early termination | -1.50 (2.263) |

17. Secondary Outcome: Change From Baseline in Lipids (Total Cholesterol [TC], Triglycerides [TG], High Density Lipoprotein Cholesterol [HDLc] and Low Density Lipoprotein Cholesterol [LDLc])
Description: Blood samples for analysis of fasting levels of lipid panel (TC, TG, HDLc and LDLc) was collected up to end of treatment or early termination. Baseline acute was Day 1 and Baseline chronic was Day 21. Change from Baseline was post-Baseline values minus Baseline values.
Time Frame: Baseline (Day 1) to Day 39
Population: Pharmacodynamic population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles/Liter (MMOL/L)
Arm/Group | GSK1278863 | Placebo
Number analyzed (Participants) | 26 | 20
Millimoles/Liter (MMOL/L)
  TC: End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  TC: End of treatment, Pre-dose | -0.69 (0.707) | 0.20 (0.689)
  TC: Early termination: number analyzed (Participants) | 2 | 0
  TC: Early termination | -0.48 (0.460) |
  TG: End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  TG: End of treatment, Pre-dose | 0.02 (0.835) | 0.27 (0.926)
  TG: Early termination: number analyzed (Participants) | 2 | 0
  TG: Early termination | -0.52 (1.160) |
  HDLc: End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  HDLc: End of treatment, Pre-dose | -0.17 (0.195) | -0.04 (0.173)
  HDLc: Early termination: number analyzed (Participants) | 2 | 0
  HDLc: Early termination | 0.13 (0.177) |
  LDLc: End of treatment, Pre-dose: number analyzed (Participants) | 21 | 18
  LDLc: End of treatment, Pre-dose | -0.53 (0.489) | 0.12 (0.701)
  LDLc: Early termination: number analyzed (Participants) | 2 | 0
  LDLc: Early termination | -0.37 (0.106) |

18. Secondary Outcome: Derived Plasma GSK1278863 Pharmacokinetic Parameter- Maximum Plasma Concentration (Cmax) and Trough Concentration (Ctau)
Description: Blood samples for pharmacokinetic analysis of GSK1278863 and selected metabolites were collected at the following time points: Visit 2-Baseline acute: pre-dose, 1 hour, 2 hours and 3.5 hours post-dose, Visit 3-post acute, Visit 4-rescreen, Visit 5-Baseline chronic and end of treatment or early termination. The actual date and time of each blood sample collection was recorded.
Time Frame: Visit 2 (Day 1): pre-dose, 1 hour, 2 hours and 3.5 hours post-dose, Visit 3 (Day 2)-post acute, Visit 4 (Day 16)-rescreen, Visit 5 (Day 23)-Baseline chronic and end of treatment (14 days after Visit 5) or early termination (between Visit 2 and 6)
Population: Pharmacokinetic concentration population comprised of all participants from whom a pharmacokinetic sample had been obtained and analyzed. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | GSK1278863 300 mg | GSK1278863 15 mg
Number analyzed (Participants) | 26 | 23
Nanogram/milliliter (ng/mL)
  Cmax: number analyzed (Participants) | 24 | 19
  Cmax | 3416.37 (81.4) | 197.28 (80.6)
  Ctau: number analyzed (Participants) | 22 | 2
  Ctau | 6.672 (131.8) | 1.357 (19.9)

19. Secondary Outcome: Derived Plasma GSK1278863 Pharmacokinetic Parameter -Area Under the Curve (AUC [0-t])
Description: as for outcome 18
Time Frame: as for outcome 18
Population: Pharmacokinetic concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram x hour/milliliter (ng*h/mL)
Arm/Group | GSK1278863 300 mg | GSK1278863 15 mg
Number analyzed (Participants) | 23 | 18
Nanogram x hour/milliliter (ng*h/mL) | 13059.70 (72.4) | 383.81 (112.2)

20. Secondary Outcome: Derived Plasma GSK1278863 Pharmacokinetic Parameter - Time to Maximum Plasma Concentration (T-max) and Last Time Point Where the Concentration is Above the Limit of Quantification (T-last)
Description: as for outcome 18
Time Frame: as for outcome 18
Population: Pharmacokinetic concentration population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK1278863 300 mg | GSK1278863 15 mg
Number analyzed (Participants) | 26 | 23
Hour
  Tmax: number analyzed (Participants) | 24 | 19
  Tmax | 1.016 [0.850 to 3.667] | 1.000 [0.833 to 3.583]
  Tlast: number analyzed (Participants) | 23 | 18
  Tlast | 22.417 [3.42 to 24.47] | 3.500 [3.37 to 23.08]

21. Secondary Outcome: Relationship of Pharmacokinetic Parameters to the Pharmacodynamic Assessments Performed in This Study
Description: A formal pharmacokinetic /pharmacodynamic analysis and pharmacokinetic /pharmacodynamic modelling for exposure relationships to endpoints was planned. The data for this outcome was not collected.
Time Frame: as for outcome 18
Population: The data for this outcome measure was not collected.
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 67 days.
Description: SAE and non-SAE were reported for the Safety population.
Groups:
- Placebo Matched With GSK1278863 15 mg: Eligible participants received placebo matched with 15 mg GSK1278863 tablets orally for 14 days.
Arm/Group | GSK1278863 300 mg | Placebo Matched With GSK1278863 300 mg | GSK1278863 15 mg | Placebo Matched With GSK1278863 15 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/20 | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/20 | 0/23 | 1/19
Other Adverse Events (participants affected / at risk) | 10/26 | 6/20 | 3/23 | 3/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 300 mg (N=26) | Placebo Matched With GSK1278863 300 mg (N=20) | GSK1278863 15 mg (N=23) | Placebo Matched With GSK1278863 15 mg (N=19)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1278863 300 mg (N=26) | Placebo Matched With GSK1278863 300 mg (N=20) | GSK1278863 15 mg (N=23) | Placebo Matched With GSK1278863 15 mg (N=19)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.